CLINICAL TRIAL: NCT06140693
Title: A Comparison of Affective Responses During Continuous and Interval Exercise
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Responsible Party: Principal Investigator, Niels Vollaard, Principal Investigator, University of Stirling
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14849
Record Dates: First submitted 2023-11-09; First posted 2023-11-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Health Behavior
Keywords: Affective valence; Exercise enjoyment
MeSH Terms: conditions — Health Behavior | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): All participants will perform all 5 exercise protocols (reduced-exertion high-intensity exercise, sprint interval exercise, below ventilatory threshold continuous exercise, at ventilatory threshold continuous exercise, and above ventilatory threshold continuous exercise) to determine the effect of intensity and duration of exercise on affective valence and felt-arousal, which will be measured using the feeling scale and felt-arousal scale respectively. Remembered enjoyment will be recorded using the physical activity enjoyment scale (PACES) 10 min post exercise.
  Interventions: Other: Continuous exercise at an intensity below the ventilatory threshold; Other: Continuous exercise at an intensity at the ventilatory threshold; Other: Continuous exercise at an intensity above the ventilatory threshold; Other: Sprint interval training; Other: Reduced-exertion high-intensity interval training

INTERVENTIONS:
Other: Continuous exercise at an intensity below the ventilatory threshold — 30 minutes of cycling exercise on a stationary bike at an intensity corresponding to 80% of the intensity at the ventilatory threshold
  Other Names: Exercise duration
Other: Continuous exercise at an intensity at the ventilatory threshold — 30 minutes of cycling exercise on a stationary bike at an intensity corresponding to 100% of the intensity at the ventilatory threshold
Other: Continuous exercise at an intensity above the ventilatory threshold — 30 minutes of cycling exercise on a stationary bike at an intensity corresponding to 110% of the intensity at the ventilatory threshold
Other: Sprint interval training — 22 min of cycling exercise on a stationary bike with a warm-up at a resistance of 25 W, followed by four 30-s 'all-out' sprints, each with a 4-min recovery intervals at 25 W
  Other Names: SIT
Other: Reduced-exertion high-intensity interval training — 10 min of cycling exercise on a stationary bike with a warm-up at a resistance of 25 W, followed by two 20-s 'all-out' sprints, with a 3-min and a 4-min recovery interval at 25 W after the first and second sprint respectively
  Other Names: REHIT

SUMMARY:
Regular exercise is important for good health, but many people do not achieve the minimum physical activity recommendations. How exercise makes people feel is an important factor in how much exercise people do. Affective valence (AV) is a measure of the pleasure and/or displeasure people feel. It has been suggested that if the drop in AV with exercise can be minimised, then people will be more likely to enjoy the exercise, and adhere to the exercise long-term.

Much research has been done to elucidate the factors that affect changes in AV with exercise, with a focus on exercise intensity. It has been hypothesised that AV will increase with low to moderate exercise intensities, but will decrease with higher exercise intensities. This has led a number of researchers to claim that there is little value in research examining the health benefits of high-intensity interval training (HIIT) and/or sprint interval training (SIT), as the exercise intensities used in these exercise routines are so high that affective valence is expected to drop to levels that are suggested to be unpalatable to members of the general public.

However, this hypothesis ignores the likely moderating effect of exercise duration: most available evidence indicates that affect drops over time with increasing exercise duration. This means that it is possible for a longer exercise bout at a lower intensity to be associated with a greater drop in AV compared to a shorter bout of exercise at a higher intensity. This may explain why recent studies have demonstrated that low-volume SIT protocols may be associated with a similar drop in AV compared to moderate-intensity continuous exercise, but are considered more enjoyable.

It is hypothesised that exercise enjoyment (and subsequent uptake and adherence to an exercise routine) is linked to the amount of time spent at reduced AV, rather than the absolute drop in AV per se. To investigate this hypothesis, changes in affective valence will be measured in response to three bouts of moderate intensity continuous exercise at different intensities but equal duration (30 minutes) as well as two bouts of SIT involving different numbers of sprint repetitions and sprint duration but equal intensity. It will be determined whether exercise enjoyment is related to the time spent at reduced levels of AV.

The overall aim of this study is to further elucidate the exercise protocol parameters that influence changes in AV with exercise.

DETAILED DESCRIPTION:
Participants:

The aim is to recruit up to 30 healthy participants (~15 men and ~15 women) from one site (University of Stirling). Participants will be reimbursed £50 for the time required to participate in this study. The required data to perform a power analysis was not available, so the number of participants will be replicated from Ekkekakis et al (2008). Exclusion criteria will be age <18 or >40 y, answering yes to one or more questions of the physical activity readiness questionnaire (PAR-Q), a resting heart rate ≥100 bpm, and/or clinically significant hypertension (>140/90 mm Hg). Blood pressure results will be provided to the participants with a note that they should contact their GP if they have any concerns about their blood pressure. Participants will be asked to visit the lab 8 times. Pregnant participants will be excluded from participation. Participants will be asked to provide written informed consent prior to participation.

Initial visit:

At least 48 hours after having been sent an electronic copy of the participant information sheet, volunteers are asked to visit our lab. The study will be fully explained, and volunteers will have the opportunity to ask any questions they may have before they are asked to sign an informed consent form. Following this, eligibility to participate will be checked by measuring height, body mass, resting blood pressure (systolic/diastolic), and heart rate, as well as current physical activity level (International Physical Activity Questionnaire; IPAQ), and potential health-related reasons why participation would not be appropriate (PAR-Q, general health questionnaire). If the volunteer is eligible to participate, then they will be asked to complete a fitness test to measure their maximal aerobic capacity (VO2max) and determine their ventilatory threshold (VT). Participants will start cycling on a stationary bike at a low intensity (50 Watts). The intensity will increase by 1 W every 3 s until volitional exhaustion or an inability to maintain pedalling frequency of 60 RPM. Expired O2 and CO2 will be continuously measured using a COSMED breath-by-breath gas analyser. VO2 is determined as the highest value for a 15-breath rolling average of VO2. The VT is determined by the procedure described by Davis et al (1979). The procedure consists of plotting the ventilatory equivalents for oxygen (VE/VO2) and carbon dioxide (VE/VCO2) over the course of the test and identifying the point at which there is a systematic increase in VE/VCO2 without a corresponding increase in VE/VO2.

Familiarisation Session:

Participants will visit the lab once more before the experimental sessions begin. In this session they will be familiarised with the continuous exercise intensities and the SIT sprints. To familiarise for the continuous exercise, each participant will cycle on the cycle ergometer for 5 min at each of the 3 intensities while ventilatory and heart rate responses are monitored. After the initial rapid increase in oxygen update (first 2-3 min), the settings on the cycle ergometer will be adjusted to elicit the desired level of VO2 (80%, 100%, and 110% of VO2 at the VT). Between each 5-min cycle (potentially longer if multiple adjustments are required), participants will be allowed to recover for as long as necessary for their heart rate to return to within 10 bpm of the pre-exercise value. Following on from this (again after heart rate has returned to within 10 bpm of pre-exercise), participants are asked to complete two maximal sprints, both of which will be performed on a mechanically braked cycle ergometer. Participants will cycle against 25 W resistance for 1 min 40 s before completing a 20-s maximal sprint against a resistance of 7.5% of their first visit bodyweight. Once this sprint is completed, participants will continue cycling against 25 W resistance for a further 3 min and 30 s before completing a 30-s maximal sprint against a resistance of 7.5% of the participant's bodyweight. After the second sprint is finished, participants will continue cycling against 25 W resistance for a further 4 min before the session is completed.

Experimental Sessions:

Sessions 3-7 will be the experimental sessions consisting of the three continuous exercise conditions and the two SIT conditions in a randomised order so as to not introduce order effects. To further decrease the risk of bias the participants will not be told which of the 3 intensities of continuous exercise they are performing.

For the three continuous exercise protocols, the participants will be asked on arrival to complete pre-exercise self-report measures (the feeling scale (FS) for affective valence; Hardy and Rejeski, 1989; and the felt-arousal scale (FAS), Svebak and Murgatroyd, 1985). The participants will then be fitted with a heart rate monitor on their chest. Participants will warm up by cycling for 5 min at 0.5 W/kg. During the final 15 s of the warm-up, participants will be asked to rate their affective valence and felt arousal. When the warm-up is completed, the resistance of the cycle ergometer will be increased to a level that matches the selected intensity for that session. This resistance will be maintained for the following 30 min. Affective valence and felt arousal will be measured during the last 15 s of minutes 3, 6, 9, 15, 18, 21, 24, 27, and 30. Once the session is completed, participants will begin a 5-min cool-down by cycling at a 0.5 W/kg resistance. Remembered enjoyment will be recorded using the PACES questionnaire 10 min after exercise completion.

For one of the SIT sessions, participants will complete a 10-min cycling bout at 25 W resistance interspersed with two 20 s supramaximal sprints. Affective valence and felt arousal will be measured at rest pre-exercise and then 15 s before each sprint, halfway through each sprint, 15 s into each sprint, at the completion of each sprint, and then 15 s after each sprint. Affective valence and felt arousal will also be measured half-way through the low-intensity sections of the protocol, at 4:30 min, and 8:30 min, as well as at the completion of the session. Heart rate and power output will also be measured throughout the session. Remembered enjoyment will be recorded using the PACES questionnaire 10 min after exercise completion.

For the other SIT session, participants will complete a 22-min cycling bout at 25 W resistance interspersed with four 30 s sprints (including a 4 min warm-up and 4-min recovery intervals after each sprint). Affective valence and felt arousal will be measured at rest pre-exercise and then 15 s before each sprint, halfway through each sprint, 25 s into each sprint, at the completion of each sprint (4:30 min, 9 min, 13:30 min, 18 min), and then 15 s after each sprint. Affective valence and felt arousal will also be measured half-way through the low-intensity sections of the protocol (6:30 min, 11 min, 15:30 min, and 20 min) as well as at the completion of the session. Heart rate and power output will also be measured throughout the session. Remembered enjoyment will be recorded using the PACES questionnaire 10 min after exercise completion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women

Exclusion Criteria:

* Age <18 or >40 y
* Answering yes to one or more questions of the physical activity readiness questionnaire (PAR-Q)
* Resting heart rate ≥100 bpm
* Clinically significant hypertension (>140/90 mm Hg)
* Students studying Sport and Exercise Science

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Affective valence | Measured pre-exercise and 10 minutes post-exercise (all protocols), every 3 minutes during continuous exercise, and 15 seconds before, halfway, 5 seconds from end of sprint, at end of sprint, and 15 seconds after each sprint for SIT protocols.
  Measured using 'the Feeling Scale' (Hardy and Rejeski, 1989) on a scale from 5 (feeling very good) to -5 (feeling very bad).
Felt-arousal | Measured pre-exercise and 10 minutes post-exercise (all protocols), every 3 minutes during continuous exercise, and 15 seconds before, halfway, 5 seconds from end of sprint, at end of sprint, and 15 seconds after each sprint for SIT protocols.
  Measured using 'Felt-arousal Scale' (Svebak and Murgatroyd, 1985) on a scale from 1 (low arousal) to 6 (high arousal)

SECONDARY OUTCOMES:
Remembered enjoyment | Measured 10 minutes post-task for all protocols.
  Measured using the physical activity enjoyment scale (PACES; Kendzierski and DeCarlo, 1991) on a scale from 0 (no enjoyment) to 48 (very high enjoyment).

CONTACTS AND LOCATIONS:
Overall Officials: Niels Vollaard, PhD, Principal Investigator — University of Stirling
Locations (1):
- University of Stirling, Stirling, Stirlingshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No